CLINICAL TRIAL: NCT06409078
Title: Clinical Study of Repeated Transcranial Magnetic Stimulation (rTMS) for Chronic Visceral Pain in Patients With Irritable Bowel Syndrome With Diarrhea (IBS-D)
Brief Title: Repetitive Transcranial Magnetic Stimulation Attenuates Visceral Pain in Irritable Bowel Syndrome With Diarrhea
Acronym: rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Soochow University (Other)
Responsible Party: Principal Investigator, Rui Li, Chief of the Department of Gastroenterology, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024156; BE2023710 (Other Grant/Funding Number: Jiangsu Provincial Department of Science and Technology); 82470573 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Irritable Bowel Syndrome; Repetitive Transcranial Magnetic Stimulation; Chronic Visceral Pain; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- repeated transcranial magnetic stimulation group (Active Comparator): The rTMS group was given 1 Hz/s for 20 min for 2 week.
  Interventions: Device: rTMS group
- sham repetitive transcranial magnetic stimulation group (Sham Comparator): For the sham rTMS group, the coil was placed over the mPFC with the rTMS function disabled, and pre-recorded acoustic artifacts were played to mimic the auditory experience of the rTMS group.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: rTMS group — Patients with IBS-D received repetitive transcranial magnetic stimulation at 1 Hz/s for 20 minutes for 2 week.
  Other Names: transcranial magnetic stimulation
  Arms: repeated transcranial magnetic stimulation group
Device: Sham device — For the sham rTMS group, the coil was placed over the mPFC with the rTMS function disabled, and pre-recorded acoustic artifacts were played to mimic the auditory experience of the rTMS group.
  Arms: sham repetitive transcranial magnetic stimulation group

SUMMARY:
Objective: To identify a central hub of visceral pain in IBS-D and elucidate the mechanism by which repetitive transcranial magnetic stimulation (rTMS) confers analgesic effects.

Design: Combined functional magnetic resonance imaging (fMRI) with visceral sensitivity assessments were used to pinpoint hyperactive brain regions of IBS-D patients. Therefore, a clinical trial was performed to validate the therapeutic potential of rTMS in IBS-D patients.

DETAILED DESCRIPTION:
Background:Chronic visceral pain in irritable bowel syndrome with diarrhea (IBS-D) is a profound therapeutic challenge. While aberrant central processing is implicated, the key brain regions driving this visceral pain and their suitability as neuromodulatory targets remain undefined.

Methods:Participants were randomly assigned (1:1) to the sham rTMS or rTMS group using a computer-generated randomization sequence created by an independent researcher who was not involved in recruitment, treatment, or outcome assessment. Allocation concealment was ensured using sequentially numbered, opaque, sealed envelopes, which were opened only after baseline evaluations were completed.

Both participants and outcome assessors were blinded to treatment allocation. The rTMS operators were not involved in data collection or analysis. For the sham condition, the coil was positioned identically over the mPFC with magnetic output disabled, and prerecorded clicking sounds were delivered to mimic the acoustic sensation of stimulation. Participants were asked not to discuss treatment sensations with assessors. Scale raters and fMRI analysts remained blinded until all analyses were finalized.

For the nested fMRI cohort, randomization and blinding procedures were identical, with group allocation revealed only after preprocessing and statistical analysis had been completed.

ELIGIBILITY:
Inclusion criteria:1.Aged between 18 and 75 years (either sex); 2.A diagnosis of IBS-D according to the Rome IV criteria;3.Experience of Bristol stool type 6 or 7 on at least 4 days per week, with a mean abdominal pain score of ≥3 (on a 0-10 scale) during the 2-week screening period.

Exclusion criteria: 1.Inflammatory or organic gastrointestinal diseases; 2.Diabetes mellitus or hyperthyroidism; 3.History of previous anorectal, intestinal, or abdominal surgery; 4.Current use of medications known to alter gastrointestinal motility or secretion; 5.Pregnancy or lactation; 6.Metallic implants or presence of a cardiac pacemaker; 7.Noncompliance with randomized treatment allocation or demonstrated poor adherence to treatment protocols.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
IBS-symptom severity score | Assessment time points were: baseline (1 week pre-treatment), end of the 2-week treatment, and post-treatment weeks 1, 2, 4, and 8.
  The criteria were based on the IBS Symptom Severity Score (IBS-SSS), a hierarchical efficacy assessment method.The IBS-SSS consists of five entries assessing the degree of abdominal pain and discomfort, frequency of abdominal pain episodes, the degree of abdominal distension and discomfort, the degree of satisfaction with bowel habits and behaviors, and the degree of impact of intestinal symptoms on life,with a total score of 500 points. A score of 75-175 is considered mild, 176-300 is moderate, and over 300 is severe. Cure was defined as a total IBS symptom severity of less than 75; efficacy was defined as 2-level improvement in total score(e.g., symptoms improved from severe to mild); validity was defined as a 1-level improvement in tatal(e.g., symptoms improved from severe to moderate or symptoms from moderate to mild); and invalidity was defined as no improvement or deterioration in total score.

SECONDARY OUTCOMES:
anorectal manometry | Assessment time points were: baseline (1 week pre-treatment), end of the 2-week treatment, and post-treatment weeks 4 and 8.
  Anorectal manometry was performed on the subjects before and after treatment and the subjects' rectal primary sensory thresholds were recorded. Rectal initial sensory thresholds between 20-90ml were considered normal , less than 20ml was considered as sensitivity rectal sensory, and cure meant that the IBS patients had their rectal initial sensory recordings restored to between 20-90ml.

OTHER OUTCOMES:
The Visceral Sensitivity Index | Assessment time points were: baseline (1 week pre-treatment), end of the 2-week treatment, and post-treatment weeks 1, 2, 4, and 8.
  The Visceral Sensitivity Index (VSI): the questionnaire is a 15-item scale used to assess visceral sensitivity. The total score ranges from 0 to 75 points, with higher scores indicating greater visceral sensitivity.
The Bristol Stool Form Scale (BSFS) | Assessment time points were: baseline (1 week pre-treatment), end of the 2-week treatment, and post-treatment weeks 1, 2, 4, and 8.
  The Bristol Stool Form Scale (BSFS): it is adopted to assess bowel habits, with scores from 1 to 7 corresponding to stool types ranging from hardest to softest, where higher scores indicate more severe diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Li, Dr., Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No